CLINICAL TRIAL: NCT04962763
Title: Correlation of Intestinal Flora and Metabolomics in Patients With Ischemic Heart
Brief Title: Correlation of Intestinal Flora and Metabolomics in Patients With Ischemic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2021230
Record Dates: First submitted 2021-07-04; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: To Search for Biomarkers Associated With Ischemic Heart Failure; To Explore the Relationship Between Intestinal Flora and Ischemic Heart Failure
Keywords: ischemic heart failure; biomarkers; intestinal flora; metabonomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma and feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure
- Control

SUMMARY:
To provide new ideas for the treatment of patients with ischemic heart failure, this study is to search for differential metabolic markers associated with ischemic heart failure and to study the influence of fecal flora on the course of heart failure in patients with ischemic heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is the final stage of all cardiovascular diseases. Myocardial damage caused by myocardial infarction, cardiomyopathy, hemodynamic overload, inflammation, or any other cause, can result in changes in myocardial structure and function, resulting in ventricular pumping and/or diastolic dysfunction. Among them, ischemic heart disease caused by coronary artery lesions is the primary cause of heart failure, clinically known as ischemic heart failure (IHF).

More and more studies have confirmed that the structure and function of the gut and the substances in the gut play an important role in the pathogenesis of heart failure, and proposed the "gut hypothesis of heart failure". Previous studies have shown that regulation of intestinal flora and its metabolites may improve the progression of patients with heart failure to some extent, but further studies are still needed to explore whether regulation of intestinal flora can effectively delay the development of heart failure and thus improve the prognosis.

This study recruited 150 patients with ischemic heart failure and 50 healthy volunteers matched with age and sex in the heart failure group required by the researchers plan to conventional drug treatment of heart failure, but in front of the collection of serum, stool samples, the patients and healthy volunteers shall be the standard diet, work and rest, time sampling (that is, the timing acquisition participants in the early morning of 2 g feces and 2 mL fasting venous blood).Metabolic profiles of serum and stool samples from patients with ischemic heart failure and healthy volunteers were studied using LC-MS, 1H NMR and 16sRNA based metabolomics and intestinal microbiome methods to identify differential metabolic markers associated with ischemic heart failure. The feces of patients with ischemic heart failure were transplanted into model rats to investigate the regulatory effects of the feces of patients with ischemic heart failure and the feces of healthy volunteers on the structure of intestinal microflora and related metabolism of normal and model animals, so as to systematically study the influence of the fecal microflora of patients with ischemic heart failure on the course of heart failure.

ELIGIBILITY:
Heart Failure Inclusion Criteria:

1. Age ≥18;
2. A clear diagnosis of coronary heart disease;
3. NYHA cardiac function grade ≥III and/or LVEF≤40%;
4. Voluntarily signed the informed consent.

Control Inclusion Criteria:

1. The spouse of the case group;
2. Age ≥18;
3. No previous clear diagnosis of coronary heart disease;
4. The LVEF: 50 ~ 80%;
5. Voluntarily signed the informed consent.

Exclusion Criteria:

1. Have received major gastrointestinal surgery (including gallbladder and appendectomy) within 5 years;
2. Inflammatory bowel disease (IBD), including ulcerative colitis, Crohn's disease, or colitis;
3. Acute gastroenteritis;
4. Clostridium difficile (recurrent) or Helicobacter pylori infection;
5. Persistent or chronic diarrhea;
6. Chronic constipation;
7. Peptic ulcer;
8. Polyps in the stomach or intestines;
9. Gastrointestinal neoplasms;
10. Irritable bowel syndrome;
11. Acute or chronic cholecystitis, hepatitis;
12. Take or inject antibiotics and probiotics in the past 3 months
13. End-stage disease (life expectancy less than 3 months);
14. Pregnant or pregnant during follow-up;
15. Failure to give informed consent (e.g. severe cognitive impairment);
16. The patient has been enrolled in other ongoing clinical trials.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No intervention. All patients diagnosed with ischemic heart failure in the Third Hospital of Peking University received the current clinical standard treatment plan, and received clinical follow-up and questionnaire survey according to this plan.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Find a new diagnostic method for ischemic heart failure | From the end of enrollment to six months
  Identify biomarkers and differential intestinal flora associated with ischemic heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, Doctor, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided